CLINICAL TRIAL: NCT03563807
Title: Feasibility and Tolerability of Group Golf Instruction Versus Tai Chi for Patients With Moderate to Advanced Parkinson's Disease
Brief Title: Golf Instruction Versus Tai Chi for People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anne-Marie Alexandra Wills, MD, Assistant Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018P000394
Record Dates: First submitted 2018-05-08; First posted 2018-06-20 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease; Movement Disorders; Neuro-Degenerative Disease
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A blinded rater will perform the Mini-BESTest of balance before and after the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Golf (Experimental): Group golf lessons will be led by professional golf instructors.
  Interventions: Other: Golf Instruction
- Tai Chi (Active Comparator): Group Tai Chi classes led by a certified Tai Chi instructor.
  Interventions: Other: Tai Chi Class

INTERVENTIONS:
Other: Golf Instruction — Subjects will participate in two weekly hour-long golf classes. Classes will be led by professional golf instructors that will work with individuals to teach participants how to play golf. This will include stretching, individual coaching, and working with participants to maximize their golf swing.
  Arms: Golf
Other: Tai Chi Class — Tai Chi is an ancient martial art that uses meditative movement to improve strength, flexibility, and balance. Subjects will participate in two weekly hour-long Tai Chi classes.The class will be led by a certified Tai Chi instructor and consist of approximately 12 people.
  Arms: Tai Chi

SUMMARY:
The purpose of this study is to determine the feasibility and tolerability of golf instruction for participants with moderate to advanced Parkinson's disease (PD). Other forms of exercise have been shown to be beneficial for PD. Golf is a low impact sport that utilizes balance and strength. Currently, there are no data looking at the effects of golf on PD. This pilot study aims to test the effects of golf in the PD patient population, particularly its effect on balance. In this study, we will be comparing group golf instruction to group Tai Chi lessons (the gold standard balance exercise for patients with PD).

DETAILED DESCRIPTION:
Approximately, 40-50 participants with Parkinson's Disease (H&Y stage 2 to 3) will be enrolled in this study. Participants who provide informed consent will be randomized 1:1 to either group golf instruction or group Tai Chi classes. Participants will be evaluated before and after the intervention with a battery of cognitive, motor and balance assessments including the UPDRS, the Mini-BESTest of balance, and timed up and go tests. They will participate in classes twice weekly for 10 weeks which will be provided free of charge. At the end of the intervention period they will repeat the assessments. The primary outcomes of the study are feasibility and tolerability. The key secondary objectives are to measure the efficacy of golf instruction on measures of balance, risk of falls.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants with a diagnosis of Parkinson's disease by a Movement Disorders specialist, H&Y stage II-III in the "On" state treated with Parkinson's disease medications
* Participants must be capable of providing informed consent and complying with trial procedures including transportation to and from classes.
* Participants must be willing and able to participate in group exercise classes.
* Participants who are engaged in physical therapy or other exercise programs must be at a stable regimen for 60 days prior to the start of the study and must be willing to maintain their current regimen for the duration of the study.

Exclusion Criteria:

* Clinical evidence of unstable medical or psychiatric illness which would prevent them from engaging in exercise
* Participants who are already active golfers or currently active in Tai Chi would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Tolerability of group golf instruction compared to Tai Chi | Both interventions will continue for 10 weeks and subject participation rates will be recorded during this time.
  The number of participants who complete 10 weeks in the study will be measured using weekly attendance sheets. We will consider the intervention to be tolerable if the proportion of participants who withdraw consent prior to the end of the study is less than 40% with 80% confidence.

SECONDARY OUTCOMES:
Safety of group golf instruction compared to Tai Chi | Both interventions will continue for 10 weeks and any adverse events will be recorded during this time.
  The frequency of treatment-related adverse events including falls will be summarized by treatment group and system organ class by CTCAE v 4.0
Key Secondary objectives are to measure the efficacy of golf instruction compared to Tai Chi on measures of balance. | Both interventions will continue for 10 weeks. The Mini-BESTest will be performed by a blinded rater before and after the intervention period.
  The Mini-BESTest will be used to measure balance before and after the intervention. The Mini-BESTest is scored from 0-28 where lower scores are better.
Activities Specific Balance Confidence Scale | Both interventions will continue for 10 weeks. Participants will complete the questionnaire before and after the intervention period.
  This is a self-reported measure of confidence in performing various ambulatory activities without falling. The scale is out of 100

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mak MK, Wong-Yu IS, Shen X, Chung CL. Long-term effects of exercise and physical therapy in people with Parkinson disease. Nat Rev Neurol. 2017 Nov;13(11):689-703. doi: 10.1038/nrneurol.2017.128. Epub 2017 Oct 13. PMID 29027544
- [Background] Li F, Harmer P, Fitzgerald K, Eckstrom E, Stock R, Galver J, Maddalozzo G, Batya SS. Tai chi and postural stability in patients with Parkinson's disease. N Engl J Med. 2012 Feb 9;366(6):511-9. doi: 10.1056/NEJMoa1107911. PMID 22316445
- [Background] Gao KL, Hui-Chan CW, Tsang WW. Golfers have better balance control and confidence than healthy controls. Eur J Appl Physiol. 2011 Nov;111(11):2805-12. doi: 10.1007/s00421-011-1910-7. Epub 2011 Mar 17. PMID 21416145
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886